CLINICAL TRIAL: NCT02268123
Title: Correlating In Vitro Fertilization Outcomes After Euploid Blastocyst Transfer With Sperm DNA Fragmentation
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2014-05
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Male Infertility
Keywords: Male Infertility; Sperm DNA Fragmentation; Sperm Abnormality
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An aliquot semen (0.5 - 1mL) will be collected and cryopreserved for analysis for DNA Fragmentation. Two tubes of serum (approximately 20 mL) will be collected from male partner via venipuncture.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if sperm DNA fragmentation is associated with in vitro fertilization (IVF) outcomes when euploid embryos are transferred.

DETAILED DESCRIPTION:
The purpose of this study is to determine if sperm DNA fragmentation is associated with in vitro fertilization (IVF) outcomes when euploid embryos are transferred. Euploid embryos are those that have a complete set of chromosomes (46, XX or 46, XY). Sperm DNA fragmentation refers to sperm DNA that is damaged or has an altered structure. The sperm chromatin structure assay (SCSA) is a method to evaluate sperm DNA Fragmentation.

Couples will undergo a routine IVF cycle at Reproductive Medicine Associates of New Jersey. Semen specimens collected on the day of ICSI will undergo semen analysis as per routine. An aliquot of semen (0.5- 1mL) will be collected for subsequent evaluation of DNA fragmentation by the Sperm Chromatin Structure Assay (SCSA) testing at SCSA Diagnostics. All embryo biopsies will undergo CCS analysis in the genomics laboratory, Foundation for Assessment and Enhancement of Embryonic Competence.

ELIGIBILITY:
Inclusion Criteria:

* Completing first IVF/ICSI cycle at Reproductive Medicine Associates of New Jersey
* Couple undergoing CCS (Comprehensive Chromosome Screening)
* Female age 35-40 years
* Male will have to refrain from ejaculation no less than 2 days but no greater than 5 days prior semen specimen production on day of oocyte retrieval

Exclusion Criteria:

* Known genetic abnormality
* Use of sperm donation or cryopreserved sperm
* Use of Oocyte donation
* Use of gestational carrier
* Use of testicular aspiration or biopsy procedures to obtain sperm
* Presence of varicosele
* Presence of hydrosalpinges that communicate with endometrial cavity
* Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation

Ages: 35 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Couples completing their first IVF/ICSI cycle at Reproductive Medicine Associates of New Jersey utilizing CCS (Comprehensive Chromosome Screening).
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2014-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
IVF/ICSI Pregnancy Outcomes with euploid blastocyst transfer based on sperm DNA fragmentation | 28 months
  rates of fertilization, blastulation, implantation, sustained implantation, delivery and miscarriage

SECONDARY OUTCOMES:
Relationship between semen analysis parameters and sperm DNA fragmentation | 28 months
  Semen analysis parameters (total motile sperm count, Volume, Concentration, Grade 1-4 )
Correlation between sperm DNA fragmentation and embryonic aneuploidy | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, HCLD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (2):
- United States (2):
  - Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey
  - Reproductive Medicine Associates of Pennsylvania at LeHigh Valley, Allentown, Pennsylvania